CLINICAL TRIAL: NCT02271360
Title: Calcium Dobesilate Versus Cabergoline for Prevention of Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: khalid-ahmed 7
Record Dates: First submitted 2014-10-19; First posted 2014-10-22 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Infertility
Keywords: infertility ICSI OHSS Calcium Dobesilate Cabergoline
MeSH Terms: conditions — Infertility | interventions — Calcium Dobesilate; Cabergoline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): In group A, (Calcium Dobesilate group), 1 cap / 8 hs Calcium Dobesilate ( 500mg) will be given from at day of HCG injection and for 21 days.
  Interventions: Drug: Calcium Dobesilate
- group B (Active Comparator): while in group B (Cabergoline group), 1 tab/day Cabergoline(Dostinex)( 0.5 mg) will be givenat day of HCG injection and for 8 days .
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Calcium Dobesilate — 1 cap / 8 hs Calcium Dobesilate ( 500mg) will be given at day of HCG injection and for 21 days
  Other Names: doxium
  Arms: group A
Drug: Cabergoline — 1 tab/day Cabergoline( 0.5 mg) will be given at day of HCG injection and for 8 days
  Other Names: Dostinex
  Arms: group B

SUMMARY:
The purpose of this study is to compare the effect of oral Calcium Dobesilate to oral Cabergoline in the prevention of ovarian hyperstimulation syndrome (OHSS) in high-risk women underwent intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
Two hundred and twenty women at risk of ovarian hyperstimulation syndrome during ICSI cycles will be randomly scheduled into two equal groups. In group A, (Calcium Dobesilate group), 1 cap / 8 hs Doxium ( 500mg) will be given at day of HCG injection and for 21 days; while in group B (Cabergoline group), 1 tab/day Cabergoline( 0.5 mg) will be given at day of HCG injection and for 8 days.

ELIGIBILITY:
Patients enrolled in the study were infertile women undergoing ICSI with one of the following criteria: previous episodes of OHSS, polycystic ovaries (i.e., > 24 antral follicles present on baseline ultrasound examination), high AMH (> 3.0 ng/mL), large number of small follicles (8 to 12 mm) seen on ultrasound during ovarian stimulation, high s.E2 at hCG trigger (E2 >3000 pg/ml or rapidly rising s.E2), presence of > 20 follicles by ultrasound on day of retrieval or large number of oocytes retrieved (> 20).

Exclusion Criteria:

* None

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with ovarian hyperstimulation syndrome (OHSS) | weekly for eight weeks
  this will be assessed by:
  Clinically:
  Abdominal bloating Mild abdominal pain Nausea ± vomiting Oliguria Acute respiratory distress syndrome
  By ultrasound Ovarian size usually ˃8 cm Ultrasound evidence of ascites
  Laboratory Haemoconcentration haematocrit ˃45% Hypoproteinaemia

SECONDARY OUTCOMES:
pregnancy rate | 14 days after embryos transfer
  β-hCG (serum hCG test) will be checked 14 days after embryos transfer

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, MD, Study Chair — lecturer of ob/gyn; ahmed saad, MD, Principal Investigator — lecturer of ob/gyn
Locations (1):
- Benha univesity hospital, Banhā, El Qualyobia, Egypt